CLINICAL TRIAL: NCT03148054
Title: Computed Tomography with Rectal Contrast and Early Endoscopy for the Detection of Anastomotic Leaks After Left Sided Colorectal Resection. a Single Center, Prospective Trial.
Brief Title: Computed Tomography Vs. Endoscopy Study
Status: Recruiting | Type: Observational
Sponsor: Spital Limmattal Schlieren (Other)
Responsible Party: Principal Investigator, Prof Urs Zingg, Head of surgery, Spital Limmattal Schlieren
Other Study IDs: 2016-01722
Record Dates: First submitted 2017-04-16; First posted 2017-05-10 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Anastomosis; Complications; Colon Disease; Leak, Anastomotic
Keywords: Anastomosis; Colon; CT; Endoscopy; Enema; Detection leak; Anastomotic leak
MeSH Terms: conditions — Colonic Diseases; Anastomotic Leak | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Patients undergoing elective left sided colon surgery
  Interventions: Device: Computer Tomography and Endoscopy

INTERVENTIONS:
Device: Computer Tomography and Endoscopy — Pelvic CT scan with i.v. and rectal contrast (Siemens Healtheneers, Erlangen, Germany) with the following scan parameters: collimation 0.6 mm, pitch 1.2 mm, CareKV with reference 120 mAs and reference 120 kV, rotation time 0.5 sec. Portal venous phase (individually tailored contrast media injection of Xenetix 300, Guerbet GmbH) and rectal contrast (500cc: 470cc water + 30cc Telebrix® gastro, a water soluble iodinated contrast agent, Guerbet GmbH).
  Endoscopy takes 5 minutes: A gastroscope with a diameter of 10mm is used for inspection of anus, rectum, anastomosis incl. measurements (distance to dentate line, diameter of anastomosis) and distal part of colon (to rule out ischemia) during short term insufflation of the rectum with CO2. No biopsies are taken. Digital photo documentation will be provided. In case of anastomotic insufficiency: optional sedation of patient and clip closure with endoscopic OTSC (over the scope clip) system.

SUMMARY:
Patients undergoing elective surgery for left-sided colon resection are asked to participate in this study: Every patient undergoes two types of examinations (endoscopy, CT scan) on day 3, 4 or 5 postoperatively. These two procedures are subject to investigation in terms of their accuracy (sensitivity, specificity) in detection of anastomotic leaks. The patients are followed up until day 42 postoperatively. There are no other specific tests or examinations within the study. Information and informed consent are obtained preoperatively.

DETAILED DESCRIPTION:
On day 3, 4 or 5 postoperatively, all patients with colorectal resection and anastomosis will undergo a CT scan with intravenous (i.v.) and rectal contrast enema and a flexible endoscopy. Both are currently routine examinations. CT scan is performed before endoscopy because contrast enema clears the rectum and anastomotic area and no further cleaning measures are necessary. The timing of the CT scan and the endoscopy is chosen because early signs of anastomotic leak should be present and thus early therapeutic interventions before the development of peritonitis is possible. The standard treatment is not altered with the exception of the two described procedures. Due to infrastructural issues and weekends the CT scan and the endoscopy can be performed on either day (3,4,5 postoperatively).

The study is to start after Ethical approval. With a sample size of 400 patients, and an annual case load of 80-100 patients (minus drop outs of 10%), the study is planned to be finished (last patient processed) 31.12.2020. Data analysis and final processing will take another 6-8 months.

All patients with colorectal disorders planned for surgery are seen in the outpatient clinic of one the four staff surgeons performing colorectal resections. This appointment is at least 1 week before surgery. During the appointment, patients are fully informed on the disease, indication, peri- and postoperative process and risk of treatment. During this visit eligibility is analysed, and information as well as informed consent are obtained.

During the entire duration of the study, all serious adverse events (SAEs) that may be causally related to the study intervention are collected and documented in source documents. Reportable events are recorded in the case report form (CRF). Study duration encompassed the time from when the participant signs the informed consent until the last protocol-specific procedure has been completed, including a safety follow-up period.

The analysis entails tests for paired categorical (McNemar test) and continuous (Student's independent t-test, Wilcoxon test) data. Sensitivity, specificity, positive and negative predictive value and accuracy will be calculated with 95% confidence interval. The significance level is set to p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic or open left sided colorectal resection with primary anastomosis (left hemicolectomy, sigmoid resection, anterior resection, segmental resection) and subtotal colectomy with anastomosis
* Male and Female patients >18 years of age
* Signed Informed Consent after being informed
* Elective surgery

Exclusion Criteria:

* Formation of a stoma during the initial operation
* For i.v. contrast CT scan: creatinine > 110 umol/l and/or glomerular filtration rate GFR < 45 ml/min, measured in the standard blood test on postoperative day 2
* Women who are pregnant. Women of childbearing age are regularly tested for possible pregnancy. Pregnancy tests are performed in the hospital at no charge
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with an investigational drug within the 30 days preceding and during the present study
* Emergency intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population entails all patients undergoing a colorectal left sided resection at the Spital Limmattal, Zurich, Switzerland according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-02-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of anastomotic leaks after left sided colon resection by Endoscopy | On postoperative day 4
  Sensitivity, specificity, positive and negative predictive value and accuracy of the diagnosis of anastomotic leak with endoscopy.

SECONDARY OUTCOMES:
Diagnosis of anastomotic leaks after left sided colon resection by Computer Tomography | On postoperative day 4
  Comparison of sensitivity, specificity, positive and negative predictive value and accuracy of the diagnosis of Anastomotic Leak of endoscopy and pelvic CT scan with rectal contrast.

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, Prof. Dr. med., Principal Investigator — Head of department (surgery)
Locations (1):
- Spital Limmattal, Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kingham TP, Pachter HL. Colonic anastomotic leak: risk factors, diagnosis, and treatment. J Am Coll Surg. 2009 Feb;208(2):269-78. doi: 10.1016/j.jamcollsurg.2008.10.015. Epub 2008 Dec 4. No abstract available. PMID 19228539
- [Background] Bakker IS, Grossmann I, Henneman D, Havenga K, Wiggers T. Risk factors for anastomotic leakage and leak-related mortality after colonic cancer surgery in a nationwide audit. Br J Surg. 2014 Mar;101(4):424-32; discussion 432. doi: 10.1002/bjs.9395. PMID 24536013
- [Background] Karliczek A, Harlaar NJ, Zeebregts CJ, Wiggers T, Baas PC, van Dam GM. Surgeons lack predictive accuracy for anastomotic leakage in gastrointestinal surgery. Int J Colorectal Dis. 2009 May;24(5):569-76. doi: 10.1007/s00384-009-0658-6. Epub 2009 Feb 17. PMID 19221768
- [Background] Facy O, Paquette B, Orry D, Binquet C, Masson D, Bouvier A, Fournel I, Charles PE, Rat P, Ortega-Deballon P; IMACORS Study. Diagnostic Accuracy of Inflammatory Markers As Early Predictors of Infection After Elective Colorectal Surgery: Results From the IMACORS Study. Ann Surg. 2016 May;263(5):961-6. doi: 10.1097/SLA.0000000000001303. PMID 26135691
- [Background] Giaccaglia V, Salvi PF, Antonelli MS, Nigri G, Pirozzi F, Casagranda B, Giacca M, Corcione F, de Manzini N, Balducci G, Ramacciato G. Procalcitonin Reveals Early Dehiscence in Colorectal Surgery: The PREDICS Study. Ann Surg. 2016 May;263(5):967-72. doi: 10.1097/SLA.0000000000001365. PMID 26528879
- [Background] Hirst NA, Tiernan JP, Millner PA, Jayne DG. Systematic review of methods to predict and detect anastomotic leakage in colorectal surgery. Colorectal Dis. 2014 Feb;16(2):95-109. doi: 10.1111/codi.12411. PMID 23992097
- [Background] Li VK, Wexner SD, Pulido N, Wang H, Jin HY, Weiss EG, Nogeuras JJ, Sands DR. Use of routine intraoperative endoscopy in elective laparoscopic colorectal surgery: can it further avoid anastomotic failure? Surg Endosc. 2009 Nov;23(11):2459-65. doi: 10.1007/s00464-009-0416-4. Epub 2009 Mar 20. PMID 19301071
- [Background] Shamiyeh A, Szabo K, Ulf Wayand W, Zehetner J. Intraoperative endoscopy for the assessment of circular-stapled anastomosis in laparoscopic colon surgery. Surg Laparosc Endosc Percutan Tech. 2012 Feb;22(1):65-7. doi: 10.1097/SLE.0b013e3182401e20. PMID 22318063
- [Background] Aryaie AH, Singer JL, Fayezizadeh M, Lash J, Marks JM. Efficacy of endoscopic management of leak after foregut surgery with endoscopic covered self-expanding metal stents (SEMS). Surg Endosc. 2017 Feb;31(2):612-617. doi: 10.1007/s00464-016-5005-8. Epub 2016 Jun 17. PMID 27317034
- [Background] Blumetti J, Abcarian H. Management of low colorectal anastomotic leak: Preserving the anastomosis. World J Gastrointest Surg. 2015 Dec 27;7(12):378-83. doi: 10.4240/wjgs.v7.i12.378. PMID 26730283
- [Background] Kornmann VN, Treskes N, Hoonhout LH, Bollen TL, van Ramshorst B, Boerma D. Systematic review on the value of CT scanning in the diagnosis of anastomotic leakage after colorectal surgery. Int J Colorectal Dis. 2013 Apr;28(4):437-45. doi: 10.1007/s00384-012-1623-3. Epub 2012 Dec 14. PMID 23239374
- [Background] Kornmann VN, van Ramshorst B, Smits AB, Bollen TL, Boerma D. Beware of false-negative CT scan for anastomotic leakage after colonic surgery. Int J Colorectal Dis. 2014 Apr;29(4):445-51. doi: 10.1007/s00384-013-1815-5. Epub 2013 Dec 20. PMID 24356897